CLINICAL TRIAL: NCT03858361
Title: Patient Specific Optimized Therapy (PSOT) in Atrial Flutter Population Miami Cardiac & Vascular Institute (MCVI) Post Marketing Surveillance (PMS) Study
Brief Title: Patient Specific Optimized Therapy (PSOT)
Acronym: PSOT
Status: Terminated | Type: Observational
Why Stopped: Philips decided to wind down the EPD Solution business
Sponsor: EPD Solutions, A Philips Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-KODEX-0011
Record Dates: First submitted 2019-02-20; First posted 2019-02-28 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Atrial Flutter Ablation — Catheter-based electrophysiological (EP) intervention.

SUMMARY:
Data collection from atrial flutter patients before, during and after undergoing catheter-based electrophysiological (EP) intervention in order to develop a patient specific optimized therapy (PSOT) to improve specific patient's arrhythmia treatment for Atrial Flutter.

DETAILED DESCRIPTION:
Prospective, single-center, non-randomized, open label, single arm study. Consented subjects who are scheduled to undergo ablation due to atrial flutter will be enrolled in the study. Data will be collected from all subjects during the ablation procedure and post procedure for a period of 3 months.

KODEX - EPD™ system will be used in all procedures during treatment of cardiac arrhythmias.

Anonymized data will be stored in an EPD database and will be used to train and test predictors for personalized optimized therapy.

Data will be collected on paper and/or electronic forms and saved in the EPD Database.

Advanced data analysis will be used to map patient specific demographics, history, current ailment, intervention to patient outcome. The technology to be utilized will help develop a method to identify the personalized treatment for a given patient (defined by: patient's demographic, history, current ailment and intervention information to achieve optimal outcome).

Data will be anonymized by removing patient protected health information, only initials will be used. The data will be integrated to an EPD data base and will be used to train and test predictors for personalized optimized therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject signed a written Informed Consent form to participate in the study, prior to any study related procedures.
* Subject is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.
* A female subject is eligible if not of child bearing potential or has a negative pregnancy test within the previous 7 days.
* Subject is deemed amenable to therapeutic ablation for atrial flutter.

Exclusion Criteria:

* Any planned surgical or endovascular intervention within 30 days before or after the index procedure.
* Subject is enrolled in another drug or device study protocol that has not reached its primary endpoint.
* Patient had experienced previous stroke (TIA or CVA).
* Thrombi detected in the heart.
* Known marked valvar insufficiency.
* Life expectancy less than 12 months.
* Known severe renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arrhythmia patients with Atrial Flutter indicated for EP procedures.
Sampling Method: Non-Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Arrhythmia recurrence The number of Arrhythmia recurrence | 3 months
  The number of arrhythmia recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Baptist Health South Florida, Florida City, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided